# **Cover Page**

Release Date: September 12, 2025

ClinicalTrials.gov ID: NCT07182838

**Unique Protocol ID:** IND 179135 Research

**Brief Title:** Proof-of-Concept Clinical Pharmacology Trial for HIV Antigen Presentation

Therapeutic Biologic Mix (HIVGP-BCG)

Official Title: Conducting an Initial Small, Controlled Clinical Pharmacology Trial to Assess for

Therapeutic Biologics Activity (Proof-of-Concept) that Suggests the Potential

for Clinical Benefits of HIV (+) Patients

**Secondary IDs:** FWA00015357 [Registry ID: DHHS, OHRP]

IRB00009424 [Registry ID: IRB, DHHS] IORG0007849 [Registry ID: IORG, DHHS]

NPI-1831468511 [Registry ID: HHS, Health Care Provider Individual] NPI-1023387701 [Registry ID: HHS, Health Care Provider Organization]

IND 179135 [Registry ID: IND, FDA]

Human APCs treat HIV antigen into small fragments, and then clear HIV virus in vivo.

# **Contents**

| 21 | CFR§ | §312.23 (a)(6) |
|---|---|---|
| Pro | tocol | <i>ls</i> 2 |
| a<br>d<br>t<br>c | ubmit<br>nd mo<br>t prov<br>escrip<br>o be u<br>ritical<br>xperir | protocol for each planned study. (Protocols for studies not submitted initially in the IND should be ited in accordance with § 312.30(a).) In general, protocols for Phase 1 studies may be less detailed one flexible than protocols for Phase 2 and 3 studies. Phase 1 protocols should be directed primarily viding an outline of the investigation - an estimate of the number of patients to be involved, a ption of safety exclusions, and a description of the dosing plan including duration, dose, or method used in determining dose - and should specify in detail only those elements of the study that are to safety, such as necessary monitoring of vital signs and blood chemistries. Modifications of the mental design of Phase 1 studies that do not affect critical safety assessments are required to be ded to FDA only in the annual report |
| p<br>t<br>a<br>e | (ii) In Phases 2 and 3, detailed protocols describing all aspects of the study should be submitted protocol for a Phase 2 or 3 investigation should be designed in such a way that, if the sponsor anticipy that some deviation from the study design may become necessary as the investigation progregalternatives or contingencies to provide for such deviation are built into the protocols at the outset example, a protocol for a controlled short-term study might include a plan for an early crossove nonresponders to an alternative therapy. | |
| • | ii)<br>rotoc | A protocol is required to contain the following, with the specific elements and detail of the olderling the above distinctions depending on the phase of study: |
| | (a) | A statement of the objectives and purpose of the study |
| | unde | The name and address and a statement of the qualifications (curriculum vitae or other statement of fications) of each investigator, and the name of each sub-investigator (e.g., research fellow, resident) working or the supervision of the investigator; the name and address of the research facilities to be used; and the name address of each reviewing Institutional Review Board. |
| | (c)<br>patie | The criteria for patient selection and for exclusion of patients and an estimate of the number of ents to be studied9 |
| | (d)<br>of me | A description of the design of the study, including the kind of control group to be used, if any, and a description ethods to be used to minimize bias on the part of subjects, investigators, and analysts9 |
| | (e)<br>dura | The method for determining the dose(s) to be administered, the planned maximum dosage, and the tion of individual patient exposure to the drug |
| | (f) | A description of the observations and measurements to be made to fulfill the objectives of the study 12 |
| | (g)<br>effec | A description of clinical procedures, laboratory tests, or other measures to be taken to monitor the ets of the drug in human subjects and to minimize risk |

It is my <u>commitment</u> that our Institutional Review Board (IRB) (IRB00009424) that complies with the requirements set forth in part 56 will be responsible for the initial and continuing review and approval of each of the studies in my proposed clinical investigation and that the sponsor-investigator (me i.e. Han Xu, M.D., Ph.D.) will report to our IRB (IRB00009424) the proposed changes in my research activity in accordance with the requirements of part 56.

I write the <u>statement</u> with respect to each clinical study involving human subjects that it either will be conducted in compliance with the institutional review board regulations in part 56 or will not be subject to the regulations under §56.104 or §56.105; and that it either will be conducted in compliance with the informed consent regulations in part 50 or will not be subject to the regulations under §50.23 and §50.24.

#### 21 CFR§312.23 (a)(6)

#### Protocols.

(i) A protocol for each planned study. (Protocols for studies not submitted initially in the IND should be submitted in accordance with § 312.30(a).) In general, protocols for Phase 1 studies may be less detailed and more flexible than protocols for Phase 2 and 3 studies. Phase 1 protocols should be directed primarily at providing an outline of the investigation - an estimate of the number of patients to be involved, a description of safety exclusions, and a description of the dosing plan including duration, dose, or method to be used in determining dose - and should specify in detail only those elements of the study that are critical to safety, such as necessary monitoring of vital signs and blood chemistries. Modifications of the experimental design of Phase 1 studies that do not affect critical safety assessments are required to be reported to FDA only in the annual report.

# The protocol for the planned IND 179135 Phase 1 clinical study NCT07182838:

In general, protocols for Phase 1 studies may be less detailed and more flexible. Phase 1 protocol of the planned IND 179135 clinical study NCT07182838 will be directed primarily at providing an outline of the clinical investigation NCT07182838 as follows:

#### > An estimate of the number of patients to be involved:

♦ 20 HIV-1 Infection Patients with controlled cancers

#### > A description of participant inclusions:

- ♦ Positive testing HIV-1 by standard PCR assay
- ♦ HIV-1 infection without symptoms
- ♦ TB negative participant is negative IGRA blood test with TB antigens.

#### > A description of safety exclusions:

- ♦ Pregnant
- ♦ Thrombosis
- ♦ Allergy
- → TB positive participant is positive IGRA blood test with TB antigens.
- ♦ AIDS Symptoms.
- ♦ Clinical signs suggestive of other infection
- ♦ Symptoms suggestive of other infection
- ♦ Evidence of critical illness

#### > A description of the dosing plan:

- ♦ Duration: 4-weeks = 28-days
- **♦** Dose:
  - 0.1 mg x 1mL HIV-1 gp160 Protein https://www.antibodies-online.com/ HIV-1 gp160 Protein Catalog No. ABIN1111556 0.1 mg x 1mL ANTIBODIES-ONLINE INC.
  - <u>Before 5 minutes</u> for the percutaneous route with the multiple puncture device, above biologic will be added into following biologic:
  - 1 Dose i.e., 50 mg wet weight organism i.e., 1 Intact Vial of lyophilized powder as follows: https://dailymed.nlm.nih.gov/dailymed/

**LABEL: BCG VACCINE** - bacillus calmette-guerin substrain tice live antigen injection, powder, lyophilized, for solution **NDC** 0052-0603-02

**BLA** 103050

Packager: Merck Sharp & Dohme Corp.

Active Ingredient(s) and Strength(s) like as following:

BCG VACCINE contains live bacteria. BCG VACCINE for percutaneous use is an attenuated, live culture preparation of the Bacillus of Calmette and Guerin (BCG) strain of Mycobacterium bovis. The TICE® strain used in this BCG VACCINE preparation. The TICE® BCG organism is grown for preparation of freeze-dried cake.

- ✓ Bacillus of Calmette and Guerin (BCG) strain of Mycobacterium bovis
- √ 1 to 8 × 10^8 colony forming units (CFU) of BCG (equivalent to approximately 50 mg wet weight)
- ✓ Merck TICE® BCG organism 50 MG wet weight
- **♦** The method to be used in determining dose:
- ♦ Purchased below FDA approved biological products according to labels:
  - 0.1 mg x 1mL HIV-1 gp160 Protein

https://www.antibodies-online.com/

HIV-1 gp160 Protein

Catalog No. ABIN1111556

0.1 mg x 1mL

ANTIBODIES-ONLINE INC.

- Before 5 minutes for the percutaneous route with the multiple puncture device, above biologic will be added into following biologic:
- 1 Dose i.e., 50 mg wet weight organism i.e., 1 Intact Vial of lyophilized powder as follows: <a href="https://dailymed.nlm.nih.gov/dailymed/">https://dailymed.nlm.nih.gov/dailymed/</a>

**LABEL: BCG VACCINE** - bacillus calmette-guerin substrain tice live antigen injection, powder, lyophilized, for solution

NDC 0052-0603-02

**BLA** 103050

Packager: Merck Sharp & Dohme Corp.

- We will specify in detail only those elements of the IND 179135 Phase 1 clinical study NCT07182838 that are critical to safety, such as necessary monitoring of vital signs and blood chemistries.
  - The vital signs of safety exclusions:
    - ✓ Pregnant
    - ✓ Thrombosis
    - ✓ Allergy
    - ✓ AIDS
    - ✓ TB positive participant is positive IGRA blood test with TB antigens.
    - ✓ Evidence of critical illness
- ♦ Modifications of the experimental design of Phase 1 studies that do not affect critical safety assessments are required to be reported to FDA only in the annual report.

#### 21 CFR § 312.30

- (a) *New protocol.* Whenever a sponsor intends to conduct a study that is not covered by a protocol already contained in the IND, the sponsor shall submit to FDA a protocol amendment containing the protocol for the study. Such study may begin provided two conditions are met:
  - (1) The sponsor has submitted the protocol to FDA for its review; and
  - (2) the protocol has been approved by the Institutional Review Board (IRB) with responsibility for review and approval of the study in accordance with the requirements of part 56. The sponsor may comply with these two conditions in either order.

Phase 1 protocols will be directed primarily at providing an outline of the investigation:

- An estimate of the number of patients to be involved:
  - ✓ 20 HIV-1 Infection Patients with controlled cancers
- A description of safety exclusions:
  - ✓ Pregnant
  - ✓ Thrombosis
  - ✓ Allergy
  - ✓ TB positive participant is positive IGRA blood test with TB antigens.
  - ✓ AIDS Symptoms.
  - ✓ Clinical signs suggestive of other infection
  - ✓ Symptoms suggestive of other infection
  - ✓ Evidence of critical illness
- A description of the dosing plan for duration:
  - ✓ Our trial duration will be 4-week duration.
- A description of the dosing plan for dose:
  - ✓ HIV-1 GP160 0.1 mg x 1.0 mL plus BCG Vaccine 50 MG Mix
- A description of the dosing plan for method to be used in determining dose:
  - ✓ HIV-1 gp160 Protein

Catalog No. ABIN1111556

0.1 mg x 1mL

ANTIBODIES-ONLINE INC.

- Before 5 minutes for the percutaneous route with the multiple puncture device, above biologic will be added into following biologic:
- ✓ LABEL: BCG VACCINE bacillus calmette-guerin substrain tice live antigen injection, powder, lyophilized, for solution

NDC 0052-0603-02

**BLA** 103050

Packager: Merck Sharp & Dohme Corp.

- The elements of the study that are critical to safety:
  - > The necessary monitoring of vital signs:
    - ✓ TB positive participant is positive IGRA blood test with TB antigens.
    - ✓ Positive testing HIV-1 by standard PCR assay.
- (ii) In Phases 2 and 3, detailed protocols describing all aspects of the study should be submitted. A protocol for a Phase 2 or 3 investigation should be designed in such a way that, if the sponsor anticipates that some deviation from the study design may become necessary as the investigation progresses, alternatives or contingencies to provide for such deviation are built into the protocols at the outset. For example, a protocol for a controlled short-term study might include a plan for an early crossover of nonresponders to an alternative therapy.

#### The IND 179135 Phase 1 clinical study need not describe Phases 2 and 3 protocols.

- (iii) A protocol is required to contain the following, with the specific elements and detail of the protocol reflecting the above distinctions depending on the phase of study:
  - (a) A statement of the objectives and purpose of the study.
  - 1. Treat Infection of Multiple HIV-1 Virus Strains.
  - 2. Activate human HIV-1 Antigen Presentation Reaction.
  - 3. The human antigen presenting cells (APCs) can treat the HIV-1 virus protein antigens into small peptide fragments, and then clear HIV-1 virus in vivo.

#### **Statement**

The objectives and purpose of the IND 179135 Phase 1 clinical study will be 2 doses of the biological product, **<u>BCG Vaccine</u>** and mix above them **before 5 minutes** to take the percutaneous use and treat the Infection of Multiple HIV-1 Virus Strains.

(b) The name and address and a statement of the qualifications (curriculum vitae or other statement of qualifications) of each investigator, and the name of each sub-investigator (e.g., research fellow, resident) working under the supervision of the investigator; the name and address of the research facilities to be used; and the name and address of each reviewing Institutional Review Board.

Contact Person: Han Xu, M.D., Ph.D., FAPCR, Sponsor-Investigator, IRB Chair, Medical Director

**Contact Company:** Medicine Invention Design Incorporation **Contact Address:** 5545 Burnside Drive, Rockville, MD 20853, USA

Contact Call: 001-301-222-7143 Contact Fax: 001-866-458-0099

Contact Email: hanxumdphd@midinc.us

# The name of investigator:

> Han Xu, M.D., Ph.D., FAPCR, Sponsor-Investigator, IRB Chair, Medical Director

Health Care Provider - Individual (NPI - 1831468511)
The address of investigator: (Online Clinical Trial Site)

> 5545 Burnside Drive, Rockville, MD 20853, USA

## The statement of the qualifications of investigator:

21 CFR 312.53(c)(1)

A signed investigator statement (Form FDA-1572) containing:

- (i) The name and address of the investigator:
  - The name of the investigator:
  - ✓ Han Xu, M.D., Ph.D., FAPCR, Sponsor-Investigator, IRB Chair, Medical Director
  - > The address of the investigator: (Online Clinical Trial Site)
  - √ 5545 Burnside Drive, Rockville, MD 20853, USA
- (ii) The name and code number, if any, of the protocol(s) in the IND identifying the study(ies) to be conducted by the investigator:
  - ✓ Han Xu, M.D., Ph.D., FAPCR, Sponsor-Investigator, IRB Chair, Medical Director
  - ✓ Health Care Provider Individual (NPI 1831468511)
  - ✓ Health Care Provider Health Maintenance Organization (Code 302R00000X)
  - ✓ IND Number: IND 179135
  - ✓ ClinicalTrials.gov ID: NCT07182838
- (iii) The name and address of any medical school, hospital, or other research facility where the clinical investigation(s) will be conducted:
  - > The name of research facility:
    - ✓ Medicine Invention Design Incorporation
    - ✓ Medicine Invention Design Incorporation (FWA00015357)
    - ✓ Medicine Invention Design Incorporation (IORG0007849)
    - ✓ Health Care Provider Group/Organization (NPI 1023387701)
    - √ Health Care Provider Health Maintenance Organization (Code 302R00000X)
    - ✓ Health Care Provider Research Clinic/Center (Code 261QR1100X)
  - The address of research facility: (Online Clinical Trial Site)
    - √ 5545 Burnside Drive, Rockville, MD 20853, USA
- (iv) The name and address of any clinical laboratory facilities to be used in the study:
  - ➤ The name of clinical laboratory facility:
    - ✓ Medicine Invention Design Incorporation
    - ✓ Medicine Invention Design Incorporation (FWA00015357)
    - ✓ Medicine Invention Design Incorporation (IORG0007849)
    - ✓ Health Care Provider Clinical Medical Laboratory (Code 291U00000X)

#### > The address of clinical laboratory facility: (Online Clinical Trial Site)

- ✓ 5545 Burnside Drive, Rockville, MD 20853, USA
- (v) The name and address of the IRB that is responsible for review and approval of the study(ies):
  - The name of the IRB:
    - ✓ Medicine Invention Design Incorporation (MIDI) IRB #1 (IRB00009424)
  - The address of the IRB: (Online Clinical Trial Site)
    - √ 5545 Burnside Drive, Rockville, MD 20853, USA
- (vi) A commitment by the investigator that he or she:
  - (a) Will conduct the study(ies) in accordance with the relevant, current protocol(s) and will only make changes in a protocol after notifying the sponsor, except when necessary to protect the safety, the rights, or welfare of subjects;
  - (b) Will comply with all requirements regarding the obligations of clinical investigators and all other pertinent requirements in this part;
  - (c) Will personally conduct or supervise the described investigation(s);
  - (d) Will inform any potential subjects that the drugs are being used for investigational purposes and will ensure that the requirements relating to obtaining informed consent (21 CFR part 50) and institutional review board review and approval (21 CFR part 56) are met:
  - (e) Will report to the sponsor adverse experiences that occur in the course of the investigation(s) in accordance with § 312.64;
  - (f) Has read and understands the information in the investigator's brochure, including the potential risks and side effects of the drug; and

#### 21 CFR 312.55(a)

Before the investigation begins, a sponsor (other than a sponsor-investigator) shall give each participating clinical investigator an investigator brochure containing the information described in § 312.23(a)(5).

(g) Will ensure that all associates, colleagues, and employees assisting in the conduct of the study(ies) are informed about their obligations in meeting the above commitments.

#### Commitment

Han Xu, M.D., Ph.D., FAPCR, Sponsor-Investigator

A commitment by the sponsor-investigator that I:

- (a) Will conduct the study (NCT07182838) in accordance with the relevant, current protocol(s) and will only make changes in a protocol after notifying the sponsor, except when necessary to protect the safety, the rights, or welfare of subjects.
- (b) Will comply with all requirements regarding the obligations of clinical investigators and all other pertinent requirements in this part.
- (c) Will personally conduct or supervise the described investigation(s).
- (d) Will inform any potential subjects that the drugs are being used for investigational purposes and will ensure that the requirements relating to obtaining informed consent (21 CFR part 50) and institutional review board review and approval (21 CFR part 56) are met;
- (e) Will report to the sponsor (Han Xu, M.D. Ph.D., FAPCR) adverse experiences that occur in the course of the investigation(s) in accordance with § 312.64.
- (f) Have read and understands the information in the investigator's brochure, including the potential risks and side effects of the drug.

#### 21 CFR 312.55(a)

Han Xu, Sponsor-Investigator, need not give an investigator brochure containing the information described in § 312.23(a)(5).

(g) Will ensure that all associates, colleagues, and employees assisting in the conduct of the study (NCT07182838) are informed about their obligations in meeting the above commitments.

(vii) A commitment by the investigator that, for an investigation subject to an institutional review requirement under part 56, an IRB that complies with the requirements of that part will be responsible for the initial and continuing review and approval of the clinical investigation and that the investigator will promptly report to the IRB all changes in the research activity and all unanticipated problems involving risks to human subjects or others, and will not make any changes in the research without IRB approval, except where necessary to eliminate apparent immediate hazards to the human subjects.

#### Commitment

Han Xu, M.D., Ph.D., FAPCR, Sponsor-Investigator, IRB Chair, Medical Director

It is my <u>commitment</u> that our Institutional Review Board (IRB) (IRB00009424) that complies with the requirements set forth in part 56 will be responsible for the initial and continuing review and approval of each of the studies in my proposed clinical investigation and that the sponsor-investigator (me i.e. Han Xu, M.D., Ph.D.) will report to our IRB (IRB00009424) the proposed changes in my research activity in accordance with the requirements of part 56.

(viii) A list of the names of the sub-investigators (e.g., research fellows, residents) who will be assisting the investigator in the conduct of the investigation(s).

## Not available right now

### The name of the research facility:

- Medicine Invention Design Incorporation (MIDI)
  - ✓ Medicine Invention Design Incorporation (FWA00015357)
  - ✓ Medicine Invention Design Incorporation (IORG0007849)
  - ✓ Health Care Provider Group/Organization (NPI 1023387701)
  - ✓ Health Care Provider Multi-Specialty Group (Code 193200000X)
  - ✓ Health Care Provider Health Maintenance Organization (Code 302R00000X)
  - √ Health Care Provider Managed Care Organization Pharmacy (Code 3336M0003X)
  - ✓ Health Care Provider Mail Order Pharmacy (Code 3336M0002X)
  - ✓ Health Care Provider Research Clinic/Center (Code 261QR1100X)
  - ✓ Health Care Provider Clinical Medical Laboratory (Code 291U00000X)

#### The address of the research facility: (Virtual / Mobile / Online)

> 5545 Burnside Drive, Rockville, MD 20853, USA

#### The name of Institutional Review Board:

- ➤ Medicine Invention Design Incorporation (MIDI) IRB #1 (IRB00009424)
- ➤ Health Care Provider Individual (NPI 1831468511)
- Health Care Provider Clinical Ethicist (Code 174V00000X)

## The address of Institutional Review Board: (Virtual / Mobile / Online)

> 5545 Burnside Drive, Rockville, MD 20853, USA

#### 21 CFR 312.53(c)(2)

**Curriculum vitae.** A curriculum vitae or other statement of qualifications of the investigator showing the education, training, and experience that qualifies the investigator as an expert in the clinical investigation of the drug for the use under investigation.

#### The statement of the qualifications of sponsor-investigator:

The education, training, and experience that qualifies the sponsor-investigator as an expert in the IND 179135 Phase 1 clinical investigation of FDA approved biological products for the use under the IND 179135 Phase 1 clinical investigation:

# The information about medical and scientific training of sponsor-investigator (SI) Han Xu, M.D., Ph.D., FAPCR, Sponsor-Investigator, IRB Chair, IORG Director

| INSTITUTION / UNIVERSITY | DEGREE /<br>TRAINING | Start Date<br>MM/YYYY | End Date<br>MM/YYYY | FIELD OF STUDY |
|---|---|---|---|---|
| Beijing Medical University (BMU)<br>School of Basic Medical Sciences (SBMS) | B.S. | 0719/86 | | Basic and Clinical<br>Medicines |
| Beijing Medical University (BMU)<br>School of Basic Medical Sciences (SBMS)<br>Department of Medicine | Internship | 09/1984 | 08/1985 | Clinical Medicines |
| Beijing Medical University (BMU)<br>School of Basic Medical Sciences (SBMS) | Internship | 09/1985 | 07/1986 | Basic Medicines |
| Beijing Friendship Hospital (BFH)<br>Beijing Clinical Research Institute (BCRI) | Residency<br>Physician | 07/1986 | 06/1991 | Internal Medicine |
| NIH-NCI accepted my degree obtained in BMU like as USA equivalent doctorate titles | M.D.<br>Ph.D. | 07/1986 | | Basic and Clinical<br>Medicines |
| National Institutes of Health (NIH)<br>National Cancer Institute (NCI) | Visiting<br>Scholar | 12/1995 | 03/2000 | Basic and Clinical<br>Research |

### The information about medical and scientific experience of sponsor-investigator (SI)

- > Han Xu, M.D., Ph.D., FAPCR, Sponsor-Investigator, IRB Chair, IORG Director
- ➤ 1980-1986 M.D., Ph.D. accepted by NIH; Beijing Medical University School of Basic Medical Science; Beijing, China

#### Dr. Han Xu received clinical education and clinical training in 1980-1986.

➤ 1986-1995 - Principal Investigator (PI), Clinical Attending Physician, Beijing Clinical Research Institute, Beijing Friendship Hospital; Beijing, China

### Dr. Han Xu received clinical training and had clinical experience in 1986-1995.

- ➤ 1995-2000 M.D., Ph.D. accepted by NIH; Visiting Scholar, NCI-Frederick, National Cancer Institute (NCI), National Institutes of Health (NIH); Frederick, Maryland
  - Dr. Han Xu received clinical investigator training in 1995-2000
- ➤ 2000-2006 Principal Investigator (PI) / Program Director (PD), Pharm1 Incorporation Beijing Office; Beijing, China
- 2006 Sponsor-Investigator (SI) / IRB Chair (Study Chair, SC) / IORG Director (Study Director, SD) / Medical Monitor (MM) / Safety Officer (SO), Medicine Invention Design Incorporation (MIDI); Rockville. Maryland
- ➤ 2013 Director Member, Medicine Invention Design Incorporation (MIDI) (IORG0007849) Institution or Organization (IORG) of Registration at U.S. Department of Health and Human Services (HHS)
- 2013 Board Member and Chair, Medicine Invention Design Incorporation (MIDI) IRB #1 (IRB00009424) Institutional Review Board (IRB) of Registration at U.S. Department of Health and Human Services (HHS) Dr. Han Xu had already been Sponsor-Investigator (SI) approved by IRB00009424.
- 2020 Active Member, Fellow of the APCR (FAPCR), Academy of Physicians in Clinical Research (APCR)
   APCR Membership Eligibility Physician Investigator
  - Certificate of Fellow of Academy of Physicians in Clinical Research (FAPCR)
  - Academy of Physicians in Clinical Research (APCR)
    - **♦ PI (Principal Investigator) in clinical trials**
    - **♦ Medical Director of Clinical Research Site**
- 2023 FDA Pre-Assignment My IND has been granted. My pre-assigned number is 179135.
  - Individual Sponsor: HAN XU
  - Organization **Sponsor**: Medicine Invention Design Incorporation
- 2023 update ClinicalTrials.gov ID: NCT07182838 under 42 CFR Part 11
  - Responsible Party (Sponsor-Investigator)
  - Study Principal Investigator [Principal Investigator (PI)]
  - Study Director (Medical Director)
  - Study Chair (IRB Chair)

- > The qualifications of sponsor-investigator:
  - ♦ Han Xu, M.D., Ph.D., FAPCR, Sponsor-Investigator, Medical Director, IRB Chair
  - ♦ NPI 1831468511 Individual
  - ♦ Clinical Ethicist (Code 174V00000X)
  - ♦ Specialist Research Study (Code 1744R1102X)
  - ♦ Pharmacist, Pharmacist Clinician (PhC) / Clinical Pharmacy Specialist (Code 1835P0018X)
  - ♦ ClinicalTrials.gov ID: NCT07182838 [Responsible Party (Sponsor-Investigator)]
  - → FWA00015357 (Human Protections Administrator)
- ➤ Medicine Invention Design Incorporation (MIDI) (IORG0007849)
- ➤ Medicine Invention Design Incorporation (MIDI) IRB #1 (IRB00009424)
- ➤ Federal-wide Assurance (FWA) for the Protection of Human Subjects (FWA00015357)
  - ♦ NPI 1023387701 Organization
  - → Multi-Specialty Group (Code 193200000X)
  - ♦ Health Maintenance Organization (Code 302R00000X)
  - → Managed Care Organization Pharmacy (Code 3336M0003X)
  - → Mail Order Pharmacy (Code 3336M0002X)
  - ♦ FDA Wholesale Drug Distributor (Maryland License Number D11379922)
  - ♦ Distribute human drug products under own label (FDA NDC Labeler Code 69891)
  - → Research Clinic/Center (Code 261QR1100X)
  - ♦ Clinical Medical Laboratory (Code 291U00000X)
- (c) The criteria for patient selection and for exclusion of patients and an estimate of the number of patients to be studied.

#### The criteria for patient selection:

- ✓ HIV-1 Infection Patients with controlled cancers
- ✓ Positive testing HIV-1 by standard PCR assay
- ✓ HIV-1 infection without symptoms
- ✓ TB negative participant is negative IGRA blood test with TB antigens.

#### The criteria for patient exclusion:

- ✓ Pregnant
- ✓ Thrombosis
- ✓ Allergy
- ✓ TB positive participant is positive IGRA blood test with TB antigens.
- ✓ AIDS Symptoms.
- ✓ Clinical signs suggestive of other infection
- ✓ Symptoms suggestive of other infection.
- ✓ Evidence of critical illness
- (d) A description of the design of the study, including the kind of control group to be used, if any, and a description of methods to be used to minimize bias on the part of subjects, investigators, and analysts.
- > Study Type: Interventional
- > Primary Purpose: Treatment
- > Study Phase: Phase 1 Clinical Trial
- > Interventional Study Model: Single Group Assignment / Single Usage / Single Dosage
- Number of Arms: 1 / single-arm study
- Masking: None (Open Label)

- > Allocation: N/A
- > Enrollment:
  - √ 20 HIV-1 Infection Patients with controlled cancers
  - ✓ Positive testing HIV-1 by standard PCR assay
  - ✓ HIV-1 infection without symptoms
  - ✓ TB negative participant is negative IGRA blood test with TB antigens.
- > Dose: HIV-1 GP160 1.0 mL plus BCG Vaccine 50 MG Mix
  - 0.1 mg x 1 mL HIV-1 GP160 as follows:

https://www.antibodies-online.com/

HIV-1 gp160 Protein

Catalog No. ABIN1111556

0.1 mg x 1mL

ANTIBODIES-ONLINE INC.

- Before 5 minutes for the percutaneous route with the multiple puncture device, above biologic will be added into following biologic:
- 1 Dose i.e., 50 mg wet weight organism i.e., 1 Intact Vial of lyophilized powder as follows:

https://dailymed.nlm.nih.gov/dailymed/

**LABEL: BCG VACCINE** - bacillus calmette-guerin substrain tice live antigen injection, powder, lyophilized, for solution

NDC 0052-0603-02

**BLA** 103050

**DLA** 103030

Packager: Merck Sharp & Dohme Corp.

- > Route: Percutaneous Use with Multiple Puncture Device
- **Duration:** Our trial duration will be 4-week duration.
- > Endpoint: Negative testing HIV-1 by standard PCR assay after percutaneous use 21 days.

# The methods to be used to minimize bias on the part of subjects, investigators, and analysts:

21 CFR 312.53(c)(1)

- (vi) A commitment by the investigator that he or she:
  - (a) Will conduct the study(ies) in accordance with the relevant, current protocol(s) and will only make changes in a protocol after notifying the sponsor, except when necessary to protect the safety, the rights, or welfare of subjects;
  - (b) Will comply with all requirements regarding the obligations of clinical investigators and all other pertinent requirements in this part;
  - (c) Will personally conduct or supervise the described investigation(s);
  - (d) Will inform any potential subjects that the drugs are being used for investigational purposes and will ensure that the requirements relating to obtaining informed consent (21 CFR part 50) and institutional review board review and approval (21 CFR part 56) are met;
  - (e) Will report to the sponsor adverse experiences that occur in the course of the investigation(s) in accordance with § 312.64;
  - (f) Has read and understands the information in the investigator's brochure, including the potential risks and side effects of the drug; and

#### 21 CFR 312.55(a)

<u>Before the investigation begins, a sponsor (other than a sponsor-investigator)</u> shall give each participating clinical investigator an investigator brochure containing the information described in § 312.23(a)(5).

(g) Will ensure that all associates, colleagues, and employees assisting in the conduct of the study(ies) are informed about their obligations in meeting the above commitments.

#### Commitment

Han Xu, M.D., Ph.D., FAPCR, Sponsor-Investigator

A commitment by the sponsor-investigator that I:

- (a) Will conduct the study (IND 179135) in accordance with the relevant, current protocol(s) and will only make changes in a protocol after notifying the sponsor, except when necessary to protect the safety, the rights, or welfare of subjects.
- (b) Will comply with all requirements regarding the obligations of clinical investigators and all other pertinent requirements in this part.
- (c) Will personally conduct or supervise the described investigation(s).
- (d) Will inform any potential subjects that the drugs are being used for investigational purposes and will ensure that the requirements relating to obtaining informed consent (21 CFR part 50) and institutional review board review and approval (21 CFR part 56) are met;
- (e) Will report to the sponsor (Han Xu, M.D. Ph.D., FAPCR) adverse experiences that occur in the course of the investigation(s) in accordance with § 312.64.
- (f) Have read and understands the information in the investigator's brochure, including the potential risks and side effects of the drug.

#### 21 CFR 312.55(a)

Han Xu, Sponsor-Investigator, need <u>not</u> give an investigator brochure containing the information described in § 312.23(a)(5).

(g) Will ensure that all associates, colleagues, and employees assisting in the conduct of the clinical study (IND 179135) are informed about their obligations in meeting the above commitments.

#### 21 CFR 312.53(c)(1)

(vii) A commitment by the investigator that, for an investigation subject to an institutional review requirement under part 56, an IRB that complies with the requirements of that part will be responsible for the initial and continuing review and approval of the clinical investigation and that the investigator will promptly report to the IRB all changes in the research activity and all unanticipated problems involving risks to human subjects or others, and will not make any changes in the research without IRB approval, except where necessary to eliminate apparent immediate hazards to the human subjects.

#### Commitment

Han Xu, M.D., Ph.D., FAPCR, Sponsor-Investigator

It is my <u>commitment</u> that our Institutional Review Board (IRB) (IRB00009424) that complies with the requirements set forth in part 56 will be responsible for the initial and continuing review and approval of each of the studies in my proposed clinical investigation and that the sponsor-investigator (me i.e. Han Xu, M.D., Ph.D.) will report to our IRB (IRB00009424) the proposed changes in my research activity in accordance with the requirements of part 56.

- (e) The method for determining the dose(s) to be administered, the planned maximum dosage, and the duration of individual patient exposure to the drug.
  - > The method for determining the single dose to be administered:
    - 0.1 mg x 1 mL HIV-1 GP160 as follows: <a href="https://www.antibodies-online.com/">https://www.antibodies-online.com/</a>
       <a href="https://www.antibodies-online.com/">https://www.antibodies-online.com/</a>
       <a href="https://www.antibodies-online.com/">https://w

- <u>Before 5 minutes</u> for the percutaneous route with the multiple puncture device, above biologic will be added into following biologic:
- 1 Dose i.e., 50 mg wet weight organism i.e., 1 Intact Vial of lyophilized powder as follows:

https://dailymed.nlm.nih.gov/dailymed/

**LABEL: BCG VACCINE** - bacillus calmette-guerin substrain tice live antigen injection, powder, lyophilized, for solution

**NDC** 0052-0603-02

**BLA** 103050

Packager: Merck Sharp & Dohme Corp.

# > The planned maximum dosage:

• 0.1 mg x 1 mL HIV-1 GP160 as follows:

https://www.antibodies-online.com/

HIV-1 gp160 Protein

Catalog No. ABIN1111556

0.1 mg x 1mL

ANTIBODIES-ONLINE INC.

- Before 5 minutes for the percutaneous route with the multiple puncture device, above biologic will be added into following biologic:
- 1 Dose i.e., 50 mg wet weight organism i.e., 1 Intact Vial of lyophilized powder as follows:

https://dailymed.nlm.nih.gov/dailymed/

**LABEL: BCG VACCINE** - bacillus calmette-guerin substrain tice live antigen injection, powder, lyophilized, for solution

**NDC** 0052-0603-02

**BLA** 103050

Packager: Merck Sharp & Dohme Corp.

Active Ingredient(s) and Strength(s) like as following:

BCG VACCINE contains live bacteria. BCG VACCINE for percutaneous use is an attenuated, live culture preparation of the Bacillus of Calmette and Guerin (BCG) strain of Mycobacterium bovis. The TICE® strain used in this BCG VACCINE preparation. The TICE® BCG organism is grown for preparation of freeze-dried cake.

- ✓ Bacillus of Calmette and Guerin (BCG) strain of Mycobacterium bovis
- ✓ 1 to 8 × 10^8 colony forming units (CFU) of BCG (equivalent to approximately 50 mg wet weight)
- ✓ Merck TICE® BCG organism 50 MG wet weight
- ➤ The duration of individual patient exposure to the drug: 4-weeks = 28-days
- **Duration:** Our trial duration will be 4-week duration.
- (f) A description of the observations and measurements to be made to fulfill the objectives of the study.
- > The observations and measurements to be made to fulfill the objectives of the study:
  - ♦ Positive testing HIV-1 by standard PCR assay before the study.
  - ♦ TB negative participant is negative IGRA blood test with TB antigens before the study.
  - ♦ Negative testing HIV-1 by standard PCR assay after 21 days of dosage
  - ♦ HIV-1 protein derivative will be positive with 1/10 Dose of HIV-1 GP160 by IGRA blood test to take the IGRA blood test with HIV-1 antigens after the percutaneous use 3 weeks of the biological product mix dosage.
- **Endpoint:** Negative testing HIV-1 by standard PCR assay after percutaneous use 21 days.

- (g) A description of clinical procedures, laboratory tests, or other measures to be taken to monitor the effects of the drug in human subjects and to minimize risk.
- ➤ Negative testing HIV-1 by standard PCR assay after percutaneous use 21 days.
- BCG should <u>not</u> be given to individuals previously infected with M. tuberculosis. A person will give the IGRA blood test with TB antigens. TB positive participant is positive IGRA blood test with TB antigens.
- ➤ BCG can activate the human antigen presenting cells (APCs) to treat HIV-1 virus target protein antigen into small peptide fragments and to clear HIV-1 virus antigens in vivo. So, the related allergen in vivo will decrease gradually.

The clinical procedures, laboratory tests, or other measures to be taken to monitor the effects of the biological product mix in human subjects and to minimize risk like as follows:

#### ➤ The clinical procedures to be taken to minimize risk:

- ✓ To take the percutaneous use can minimize risk.
- ✓ 2 doses of the biological product, <u>HIV-1 GP160</u> add into 1 dose of the biological product, <u>BCG VACCINE</u> and mix above them **before 5 minutes** to take the percutaneous use.
- ✓ BCG can activate the human antigen presenting cells (APCs) to treat HIV-1 virus target protein antigen into small peptide fragments and to clear HIV-1 virus antigens in vivo. So, the related allergen in vivo will decrease gradually.

# The clinical and laboratory tests to be taken to monitor the effects of the biological product mix in human subjects:

- ✓ Positive testing HIV-1 by standard PCR assay before the study.
- ✓ Negative testing HIV-1 by standard PCR assay after 21 days of dosage
- ✓ HIV-1 protein derivative will be positive with 1/10 Dose HIV-1 GP160 by the IGRA blood test to take the IGRA blood test with HIV-1 antigens after percutaneous use 3 weeks of the biological product mix dosage.

#### The clinical and laboratory tests to be taken to minimize risk:

- > The risk exclusions like as following:
- ♦ Pregnant
- ♦ Thrombosis
- ♦ Allergy
- ♦ TB positive participant is positive IGRA blood test with TB antigens.
- ♦ AIDS Symptoms
- ♦ Clinical signs suggestive of other infection
- ♦ Symptoms suggestive of other infection
- ♦ Evidence of critical illness

#### 21 CFR 312.10(a)

A sponsor may request FDA to waive applicable requirement under this part. A waiver request may be submitted either in an IND or in an information amendment to an IND.

### [21 CFR 312.10(a)(3)]

Other information justifying a waiver.

According to 21 CFR 312.10(a), the sponsor (Han Xu, M.D., Ph.D., FAPCR) needs to request FDA to waive applicable requirement under this part which means 21 CFR Part 312. Therefore, my investigation must waive the requirements of 21 CFR 312.53(c). In particular, my investigation must waive the requirements of 21 CFR 312.53(c)(1). Also, my clinical investigation must waive the requirements of 21 CFR §312.305 (c)(1) and 21 CFR §312.305 (c)(3). Although I am not a licensed physician, I still can be a qualified sponsor-investigator for my IND Phase I clinical investigation.

#### 21 CFR 312.53(c)(1)(vi)(d)

Will inform any potential subjects that the drugs are being used for investigational purposes and will ensure that the requirements relating to obtaining informed consent (21 CFR part 50) and institutional review board review and approval (21 CFR part 56) are met;

I write the <u>statement</u> with respect to each clinical study involving human subjects that it either will be conducted in compliance with the institutional review board regulations in part 56 or will not be subject to the regulations under §56.104 or §56.105; and that it either will be conducted in compliance with the informed consent regulations in part 50 or will not be subject to the regulations under §50.23 and §50.24.

#### 21 CFR 312.53(c)(1)(vii)

A commitment by the investigator that, for an investigation subject to an institutional review requirement under part 56, an IRB that complies with the requirements of that part will be responsible for the initial and continuing review and approval of the clinical investigation and that the investigator will promptly report to the IRB all changes in the research activity and all unanticipated problems involving risks to human subjects or others, and will not make any changes in the research without IRB approval, except where necessary to eliminate apparent immediate hazards to the human subjects.

It is my <u>commitment</u> that our Institutional Review Board (IRB) (IRB00009424) that complies with the requirements set forth in part 56 will be responsible for the initial and continuing review and approval of each of the studies in my proposed clinical investigation and that the sponsor-investigator (me i.e. Han Xu, M.D., Ph.D.) will report to our IRB (IRB00009424) the proposed changes in my research activity in accordance with the requirements of part 56.

To minimize potential bias resulting from orally verbal voice administration of assessments, the sponsor (Han Xu, M.D., Ph.D., FAPCR) will consider using automated virtual interviewers to administer the assessments remotely. According to similar principles, the formal pre-IND review will be conducted in the format -- written response only (WRO) by email.

# Han Xu, M.D., Ph.D., FAPCR, Sponsor-Investigator, Medical Director, IRB Chair, IORG Director

- > NPI 1831468511 Individual
  - Clinical Ethicist (Code 174V00000X)
  - Specialist Research Study (Code 1744R1102X)
  - Pharmacist, Pharmacist Clinician (PhC) / Clinical Pharmacy Specialist (Code 1835P0018X)
- Certificate of Fellow of Academy of Physicians in Clinical Research (FAPCR)
  - Principal Investigator (PI) in clinical trials
  - Medical Director of Clinical Research Site
- ➤ Medicine Invention Design Incorporation (MIDI) (IORG0007849) -- IORG Director (IORG0007849)
- Medicine Invention Design Incorporation (MIDI) IRB #1 (IRB00009424) -- IRB Chair (IRB00009424)
- > Federal-wide Assurance (FWA) for the Protection of Human Subjects (FWA00015357)
  - Human Subjects Administrator (FWA00015357)
- > FDA Wholesale Drug Distributor (Maryland License Number: D11379922) -- Medical Director (D11379922)
- > NPI 1023387701 Organization
  - Multi-Specialty Group (Code 193200000X)
  - Research Clinic/Center (Code 261QR1100X)
  - Clinical Medical Laboratory (Code 291U00000X)
  - Health Maintenance Organization (Code 302R00000X)
  - Managed Care Organization Pharmacy (Code 3336M0003X) -- Mail Order Pharmacy (Code 3336M0002X)
  - FDA Wholesale Drug Distributor (Maryland License Number: D11379922)
  - Distribute human drug products under own private label (FDA NDC Labeler Code 69891)
  - FDA Establishment Identifier (FEI Number 300363713)
- > FDA Pre-Assignment application My IND has been granted. My pre-assigned number is IND 179135.
  - Individual Sponsor: HAN XU
  - Organization Sponsor: Medicine Invention Design Incorporation
- ClinicalTrials.gov ID: NCT07182838 under 42 CFR Part 11
  - Responsible Party: Sponsor-Investigator: Han Xu, M.D., Ph.D., FAPCR
  - Study Principal Investigator [Principal Investigator (PI)]: Han Xu, M.D., Ph.D., FAPCR
  - Study Director (Medical Director): Han Xu, M.D., Ph.D., FAPCR
  - Study Chair (IRB Chair): Han Xu, M.D., Ph.D., FAPCR